CLINICAL TRIAL: NCT07060859
Title: The Influence of The Topical Combined Application of Dexamethasone, Ascorbic Acid, and β-Sodium Glycerophosphate on Implant Osseointegration: A Randomized Clinical Trial
Brief Title: Topical Dexamethasone, Ascorbic Acid, and BGP for Enhancing Implant Osseointegration
Acronym: DAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manar Ziad Foura-Matar (Other)
Responsible Party: Sponsor-Investigator, Manar Ziad Foura-Matar, Dentist ( Implantologist), Al-Azhar University - Gaza
Organization: Al-Azhar University - Gaza (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAG-RCT-2023
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Implant Stability and Osseointegration
Keywords: dexamethasone; ascorbic acid; β-sodium glycerophosphate; osseointegration; implant stability quotient; implant stability; resonance frequency analysis; osteogenic inducer; Immediate dental implants
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: This study followed a split-mouth design, analyzed using a parallel assignment model at the implant level. Each participant received two dental implants: one implant served as the intervention site and received a topical application of dexamethasone, ascorbic acid, and β-sodium glycerophosphate, while the other implant served as the control site and received standard placement without any topical application. Both implants were placed during the same surgical session, allowing for intra-patient comparison under identical clinical and systemic conditions. Implant stability was assessed at multiple time points using resonance frequency analysis (RFA).
Who Masked: Participant, Outcomes Assessor
Masking Description: This was a single-blind study in which participants were unaware of which implant site received the topical intervention. The care provider and investigator were aware of the allocation. Outcome assessors were masked to the assignment to ensure unbiased evaluation of implant stability measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Test) (Experimental): Participants received a dental implant with the topical application of dexamethasone, ascorbic acid, and β-sodium glycerophosphate during surgery.
  Interventions: Drug: Topical Application of Dexamethasone, Ascorbic Acid, and β-Sodium Glycerophosphate
- Control (No Intervention): Participants received a dental implant using the standard surgical procedure without any topical application.

INTERVENTIONS:
Drug: Topical Application of Dexamethasone, Ascorbic Acid, and β-Sodium Glycerophosphate — A topical combination of dexamethasone (anti-inflammatory), ascorbic acid (antioxidant), and β-sodium glycerophosphate (mineralization support) was applied directly to the implant site during surgery. The intervention aimed to enhance early osseointegration by modulating local biological responses.
  Arms: Intervention (Test)

SUMMARY:
The goal of this clinical trial was to evaluate whether the topical application of a combination of dexamethasone, ascorbic acid, and β-sodium glycerophosphate could enhance implant osseointegration in adult dental implant patients. The main question it aimed to answer was:

Did the combined topical use of these agents improve implant stability during the healing phase?

Researchers compared intervention implants (which received the topical agents at the implant site) to control implants (which received standard placement without topical application) within the same participant, in order to assess differences in implant stability and osseointegration.

Participants:

Underwent dental implant surgery.

Received both the topical treatment and the standard procedure, applied to different implant sites.

Returned for follow-up visits, where implant stability was measured using resonance frequency analysis (RFA) at predefined time intervals.

DETAILED DESCRIPTION:
This randomized clinical trial was conducted to investigate the effect of the topical application of a combination of dexamethasone, ascorbic acid, and β-sodium glycerophosphate on the osseointegration of dental implants. The rationale behind the study was based on existing evidence suggesting that these agents may enhance bone healing, reduce inflammation, and support mineralization when applied locally.

Each participant received two dental implants: one designated as the intervention site (treated with the topical combination of the three agents at the time of implant placement), and the other as the control site (placed without any topical application). This split-mouth design allowed intra-individual comparison, minimizing the influence of patient-related variability.

Implant stability was assessed using resonance frequency analysis (RFA) at four follow-up intervals to evaluate differences in osseointegration between the two sites. The study aimed to determine whether the adjunctive use of these agents could improve early implant stability, potentially contributing to more predictable outcomes in dental implantology.

No investigational drugs or devices were used beyond standard clinical tools. The study was approved by a local ethics committee, and informed consent was obtained from all participants prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Provided a written informed consent prior to initiation of any study procedures.
2. Was able to understand and agrees to comply with planned study procedures and be available for all study visits.
3. Agreed to undergo cone beam computed tomography (CBCT) imaging.
4. Was a male or non-pregnant female, >/= to 18 years of age at the time of enrollment.
5. Was in good general health, free medical diseases.
6. Had two hopeless teeth for minimum required extraction for the purpose of implant-supported restorations.

Exclusion Criteria:

1. Was undergoing chronic treatment with any medication known to affect oral status and bone turnover.
2. Had a contraindication for surgical treatment.
3. Was suffering from a known psychological disorder.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Implant Stability Measured by Implant Stability Quotient (ISQ) Using Resonance Frequency Analysis (RFA) | At baseline (day of surgery), 4 weeks, 8 weeks, and 16 weeks post-surgery
  Implant stability will be assessed using resonance frequency analysis (RFA), with results reported as Implant Stability Quotient (ISQ) values. The ISQ scale ranges from 1 (lowest stability) to 100 (highest stability). Higher ISQ values indicate better implant stability and osseointegration.

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar University - Faculty of Dentistry - Gaza, Gaza, Gaza Strip, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to confidentiality considerations and the absence of a formal data-sharing infrastructure. The study was not initially designed with data sharing in scope.